CLINICAL TRIAL: NCT02305134
Title: Tipepidine in Children With Attention Deficit/Hyperactivity Disorder (AD/HD): a Double-blind, Placebo-controlled Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chiba University (Other)
Responsible Party: Principal Investigator, Tsuyoshi Sasaki, Department of Child Psychiatry, Chiba-University Hospital, Chiba University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: G26023; UMIN000015748 (Other: UMIN Clinical Trials Registry (UMIN-CTR))
Record Dates: First submitted 2014-11-27; First posted 2014-12-02 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Attention Deficit Disorder With Hyperactivity Disease; Hyperkinesis; Attention Deficit and Disruptive Behavior Disorders
Keywords: Tipepidine, GIRK
MeSH Terms: conditions — Hyperkinesis; Attention Deficit and Disruptive Behavior Disorders | interventions — tipepidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tipepidine Hibenzate (Active Comparator): Tipepidine is taken orally at 30 mg/day (10 mg after breakfast, 10 mg after supper, and 10 mg before bedtime), for 4 weeks.
  Interventions: Drug: Tipepidine Hibenzate
- Placebo (Placebo Comparator): Placebo is taken orally after breakfast, after supper, and before for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tipepidine Hibenzate
  Arms: Tipepidine Hibenzate
Drug: Placebo
  Arms: Placebo

SUMMARY:
Tipepidine (3-[di-2-thienylmethylene]-1-methylpiperidine) has been used solely as a nonnarcotic antitussive in Japan since 1959. The safety of tipepidine in children and adults has already been established. It is reported that tipepidine inhibits G-protein-coupled inwardly rectifying potassium (GIRK)-channel currents. The inhibition of GIRK channels by tipepidine is expected to modulate the level of monoamines in the brain. We put forward the hypothesis that tipepidine can improve attention deficit/hyperactivity disorder (ADHD) symptoms by modulating monoaminergic neurotransmission through the inhibition of GIRK channels. The purpose of this double-blind, placebo-controlled trial is to confirm whether treatment with tipepidine can improve symptoms in pediatric patients with ADHD.

DETAILED DESCRIPTION:
Tipepidine (3-[di-2-thienylmethylene]-1-methylpiperidine) has been used solely as a nonnarcotic antitussive in Japan since 1959. The safety of tipepidine in children and adults has already been established. It is reported that tipepidine inhibits G-protein-coupled inwardly rectifying potassium (GIRK)-channel currents. The inhibition of GIRK channels by tipepidine is expected to modulate the level of monoamines in the brain. We put forward the hypothesis that tipepidine can improve attention deficit/hyperactivity disorder (ADHD) symptoms by modulating monoaminergic neurotransmission through the inhibition of GIRK channels. The purpose of this double-blind, placebo-controlled trial is to confirm whether treatment with tipepidine can improve symptoms in pediatric patients with ADHD.

See our previous open trial, An Open Study of Tipepidine Hibenzate in Patients With Attention Deficit Hyperactivity Disorder (ADHD) http://clinicaltrials.gov/show/NCT01835093

ELIGIBILITY:
[Inclusion Criteria]

1. Diagnosis of attention deficit hyperactivity disorder besed on DSM-5 criteria.
2. Scores of 20 or higher in ADHD-RS (physician evaluation) total score.
3. currently is an outpatient at Chiba University Hospital Department of Psychiatry or Child Psychiatry.
4. currently receiving no medications for ADHD (atomoxetine, methylphenidate) treatment for the previous 4 weeks prior to enrollment in this study.
5. currently receiving no medications of antidepressants, mood stabilizers and the antipsychotics treatment for the previous 4 weeks prior to enrollment in this study.
6. currently receiving no medications of GIRK channel antagonist (tipepidine, cloperastine, caramiphen) treatment for the previous 4 weeks prior to enrollment in this study.
7. Ages 6 - 17, male or female
8. Provision of written informed consent by patients and parents or guardian.
9. must be able to swallow capsuled medicine.

[Exclusion Criteria]

1. History of allergic reaction or hypersensitivity to tipepidine hibenzate.
2. Patients who have not been informed of having the disease at the time of informed consent.
3. Diagnosis of any of the following diseases based on the DSM-5 criteria. Autism Spectrum Disorder, Schizophrenia Spectrum and Other Psychotic Disorders, Neurocognitive Disorders, Substance Related and Addictive Disorders, Feeding and Eating Disorders, Personality Disorders, Paraphilic Disorders.
4. currently receiving medications for ADHD (atomoxetine, methylphenidate) treatment for the previous 4 weeks prior to enrollment in this study.
5. currently receiving medications of antidepressants, mood stabilizers and the antipsychotics treatment for the previous 4 weeks prior to enrollment in this study.
6. currently receiving medications of GIRK channel antagonist (tipepidine, cloperastine, caramiphen) treatment for the previous 4 weeks prior to enrollment in this study.
7. Somatic disorder which requires severe body management or severe meal management.
8. participating in another clinical trial within 3 months prior to enrollment into this study. (except for observation study without intervention).
9. planning change of treatment because of unstable neurological manifestations or somatic symptoms.
10. History of suicidal ideation within the past year.
11. pregnant or nursing, or intending to become pregnant or to start breastfeeding during the study.
12. Other clinically significant reasons for exclusion by investigators.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2015-06-11 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
The ADHD Rating Scale IV Japanese Version (ADHD-RS-IV-J) by physician. | Changes from baseline in ADHD-RS-IV-J at 4-weeks
  The ADHD Rating Scale-IV obtains parent ratings regarding the frequency of each ADHD symptom based on DSM-IV criteria. The ADHD Rating Scale-IV is completed independently by the parent and scored by a clinician. The scale consists of 2 subscales: inattention (9 items) and hyperactivity-impulsivity (9 items).

SECONDARY OUTCOMES:
Subscores (Inattentive subscore, Hyperactive/impulsive subscore) of the ADHD-RS-IV-J by physician. | Changes from baseline in at 4-weeks
Total scores and subscores (Inattentive subscore, Hyperactive/impulsive subscore) of the ADHD-RS-IV-J by parents. | Changes from baseline in at 4-weeks
Total scores and subscores (planning subscore, attention subscore, simultaneous subscore, successive subscore) of DN-CAS (Das-Naglieri Cognitive Assessment System) Japanese Version. | Changes from baseline in at 4-weeks
  The DN-CAS is an assessment battery designed to evaluate cognitive processing. It was developed to integrate theoretical and applied areas of psychological knowledge using cognitive processing theory and tests designed to measure-Planning, Attention, Simultaneous, and Successive Processing (PASS)-in individuals ages 5-17. This assessment facilitates mental health professionals in the identification of Attention-Deficit/Hyperactivity Disorder, Traumatic Brain Injury, learning disabilities, Mental Retardation, and giftedness.
Scores of CGI-ADHD-S, CGI-ADHD-I | Changes from baseline in at 4-weeks
Biologocal markers (Serum levels of Pro-BDNF, Mature-BDNF, Oxytocin) | Changes from baseline in at 4-weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, Chiba University School of Medicine, Chiba, Chuo-ku, Japan